CLINICAL TRIAL: NCT07380399
Title: Transulnar Access in Patients With Ipsilateral Radial Artery Occlusion Undergoing Coronary Angiography or Angioplasty: Safety and Effect on Hand Function (ULNART)
Brief Title: Transulnar Access in Patients With Ipsilateral Radial Artery Occlusion Undergoing Coronary Angiography or Angioplasty
Acronym: ULNART
Status: Recruiting | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Karelas Dimitrios, Principal Investigator, National and Kapodistrian University of Athens
Other Study IDs: 21171-01/12/2025
Record Dates: First submitted 2026-01-21; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Radial Artery Occlusion; Vascular Access; Coronary Artery Disease (CAD)
Keywords: Radial Artery Occlusion; Ulnar Artery; Coronary Angiography; Percutaneous Coronary Intervention; Upper Limb Function; Transulnar Access
MeSH Terms: conditions — Arterial Occlusive Diseases; Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ULNART Cohort: Adults with documented radial artery occlusion undergoing elective coronary angiography or angioplasty, in whom transulnar arterial access ipsilateral to the occluded radial artery is selected by the treating physician. Participants are followed prospectively to assess vascular safety and hand function outcomes.

SUMMARY:
Coronary angiography and angioplasty are commonly performed through the radial artery at the wrist as this approach is associated with fewer bleeding complications and faster recovery. In some patients, the radial artery becomes occluded after prior procedures, requiring selection of an alternative access site for future coronary interventions.

The ulnar artery is a potential alternative wrist access. However, limited data are available on the safety of using the ulnar artery in the same arm as an occluded radial artery and on the possible effects on hand strength, sensation, and daily hand function.

The goal of this observational study is to evaluate the safety of transulnar access and its effect on hand function in adults with ipsilateral radial artery occlusion undergoing coronary angiography or angioplasty.

The main questions addressed by the study are:

* How often do serious access-related vascular or nerve complications occur?
* Does hand strength, sensation, or functional use of the hand change during follow-up?
* Does the ulnar artery remain patent after the procedure? The choice of vascular access site is made by the treating physician based on clinical judgment. Participants who undergo transulnar access will undergo follow-up assessments, including ultrasound evaluation of arm arteries, standardized hand function testing, and short questionnaires assessing upper-limb function.

The findings of this study are expected to inform access-site selection, improve patient counseling, and support safer care for patients with radial artery occlusion undergoing coronary procedures.

DETAILED DESCRIPTION:
Transradial access is the preferred approach for coronary angiography and angioplasty because it is associated with reduced bleeding complications and faster recovery compared with femoral access. Radial artery occlusion is a recognized complication of transradial procedures and may limit future use of this access site. In patients with radial artery occlusion, selection of an alternative vascular access is required, particularly when preservation of the contralateral radial artery is clinically important.

The ulnar artery represents an anatomically plausible alternative upper-limb access route, contributing substantially to hand perfusion through the palmar arterial network. However, concerns remain regarding the vascular and functional safety of transulnar access, especially when used ipsilateral to a pre-existing radial artery occlusion. Available evidence is limited and methodologically heterogeneous, with inconsistent assessment of vascular integrity and hand function.

ULNART is a prospective observational cohort designed to evaluate the safety and functional outcomes of transulnar arterial access in patients with ipsilateral radial artery occlusion undergoing coronary angiography or angioplasty. Vascular access selection is determined by the treating physician and is not assigned by the study protocol. The study observes outcomes following transulnar access without influencing procedural decision-making.

Participants undergo standardized baseline and follow-up assessments integrating vascular imaging, objective neuromuscular testing, and patient-reported outcome measures. Color duplex ultrasonography is used to assess upper-limb arterial anatomy and ulnar artery patency, while hand function is evaluated using quantitative strength testing, sensory assessment, and validated questionnaires addressing upper-limb function and cold sensitivity. Assessments are repeated shortly after the procedure and at predefined later time points to evaluate recovery and detect early or delayed access-related effects.

The primary objective is to estimate the incidence of serious access-related vascular and clinical neuromuscular complications. Secondary objectives include characterization of ulnar artery patency, changes in hand strength and sensory function over time, patient-reported functional outcomes, and identification of factors associated with adverse events. Data are collected prospectively using standardized protocols and analyzed according to a prespecified statistical analysis plan appropriate for an observational cohort.

The results of ULNART are expected to provide systematic evidence on the vascular safety and functional impact of transulnar access in patients with radial artery occlusion, supporting informed access-site selection and patient counseling when transradial access is unavailable or clinically undesirable.

ELIGIBILITY:
Inclusion Criteria

Participants must meet all of the following criteria to be eligible:

* Adults aged 18 years or older
* Documented radial artery occlusion in the upper limb intended for vascular access, confirmed by ultrasound or angiography
* Scheduled to undergo elective coronary angiography and/or angioplasty
* Transulnar arterial access on the same side as the occluded radial artery is selected by the treating physician
* Contralateral radial artery access is not feasible or is clinically undesirable, including for reasons such as:
* documented occlusion or severe disease of the contralateral radial artery
* unfavorable anatomy or prior failed access
* strategic preservation of the contralateral radial artery for future surgical or dialysis needs
* Adequate ulnar artery flow and anatomy for access, as assessed by pre-procedural ultrasound
* Able and willing to provide written informed consent

Exclusion Criteria

Participants meeting any of the following criteria will be excluded:

* Inadequate or absent ulnar artery flow at the intended access site on ultrasound
* Known ulnar nerve injury or neuropathy affecting the access-side upper limb
* Severe pre-existing motor or sensory dysfunction of the access-side hand that would interfere with functional assessment
* Emergency coronary procedures that preclude baseline vascular or functional assessment
* Participation in another interventional clinical study involving vascular access or intervention in the same upper limb
* Local conditions at the intended access site, such as active infection, burn, or extensive scarring
* Pregnancy or breastfeeding
* Life expectancy less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants are recruited from cardiac catheterization laboratories and cardiology services of two tertiary-care public hospitals in Greece, including high-volume referral centers performing invasive coronary procedures. The study population represents adults undergoing routine elective coronary angiography or angioplasty in these hospital settings, where vascular access decisions are made as part of standard clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 127 (Estimated)
Dates: Start 2025-11-01 (Actual); Primary Completion 2030-01 (Estimated); Study Completion 2032-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Access-Related Vascular and Clinical Neuromuscular Complications | 30 days
  Composite incidence of serious vascular and clinical neuromuscular complications attributable to transulnar arterial access ipsilateral to radial artery occlusion. Serious vascular events include acute hand ischemia, symptomatic ulnar artery occlusion, flow-limiting dissection requiring treatment, pseudoaneurysm or arteriovenous fistula requiring intervention, major access-site hematoma, or major bleeding. Clinical neuromuscular events include new, clinically evident motor or sensory deficits in the ulnar nerve distribution that persist or require targeted therapy.

SECONDARY OUTCOMES:
Number of Access Attempts | During the index procedure
  Number of puncture attempts required to obtain successful vascular access
Technical Success Without Access-Site Crossover | During the index procedure
  Successful completion of coronary angiography or angioplasty via intended transulnar access without conversion to an alternative vascular access site.
Procedure Duration | During the index procedure
  Total procedural time from vascular access to sheath removal
Ulnar Artery Patency | Within 24 hours, 30 days, and 180 days
  Assessment of ulnar artery patency and flow characteristics using color duplex ultrasonography, including presence of antegrade flow and absence of occlusion or flow-limiting abnormalities.
Early Access-Related Vascular and Neuromuscular Complications | Within 24 hours after band removal
  Incidence of access-related vascular and neurologic complications occurring within 24 hours after removal of the hemostatic device, including minor bleeding, hematoma, reversible neurologic symptoms, and access-site findings not meeting criteria for the primary endpoint.
Change in Handgrip Strength | Within 24 hours, 30 days, and 180 days
  Change from baseline in handgrip strength of the access-side hand measured with a calibrated dynamometer.
Change in Key Pinch Strength | Within 24 hours, 30 days, and 180 days
  Change from baseline in key (lateral) pinch strength of the access-side hand measured with a calibrated pinch gauge.
Change in Sensory Function | Within 24 hours, 30 days, and 180 days
  Change from baseline in tactile sensation of the ulnar nerve distribution assessed using standardized light-touch threshold testing.
Change in Patient-Reported Upper-Limb Function | 10 days, 30 days and 180 days
  Change from baseline in patient-reported upper-limb function assessed using validated questionnaires evaluating disability and cold sensitivity.
Late Vascular or Neuromuscular Complications | 6 months
  Incidence of vascular or neurologic complications occurring beyond 30 days that do not meet primary endpoint criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Aznaouridis, Ass. Professor of Cardiology, Principal Investigator — 1st Department of Cardiology, Hippokration Hospital, National and Kapodistrian University of Athens; Dimitrios Karelas, MD, Principal Investigator — National and Kapodistrian University of Athens; Ioannis Tsiafoutis, MD, PhD, Principal Investigator — 2nd Department of Cardiology, Hellenic Red Cross Hospital
Locations (2):
- Greece (2):
  - Hellenic Red Cross Hospital, Athens
  - Hippokratio General Hospital, Athens

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the results reported in publications arising from this study will be made available, including demographic variables, procedural characteristics, vascular imaging findings, functional test results, and patient-reported outcome measures. A corresponding data dictionary and study protocol will be provided. Data will be shared after publication of the primary results, upon reasonable request, subject to approval by the study investigators and completion of a data-use agreement, in accordance with applicable ethical approvals and data protection regulations.
Supporting Information: Study Protocol, SAP, Analytic Code

REFERENCES:
- [Background] Roghani-Dehkordi F, Hosseinzadeh H, Kermani-Alghoraishi M, Khosravi A, Vakhshoori M, Sadeghi M, Danesh M, Sadeghi N, Sahfie D. The transulnar approach in the patients with ipsilateral radial artery occlusion. ARYA Atheroscler. 2020 Jan;16(1):33-38. doi: 10.22122/arya.v16i1.2016. PMID 32499829
- [Background] Hsueh SK, Cheng CI, Fang HY, Omran MM, Liu WH, Chung WJ, Chen CJ, Yang CH, Fang CY, Wu CJ. Feasibility and Safety of Transulnar Catheterization in Ipsilateral Radial Artery Occlusion. Int Heart J. 2017 May 31;58(3):313-319. doi: 10.1536/ihj.16-244. Epub 2017 May 12. PMID 28496021
- [Background] Kedev S, Zafirovska B, Dharma S, Petkoska D. Safety and feasibility of transulnar catheterization when ipsilateral radial access is not available. Catheter Cardiovasc Interv. 2014 Jan 1;83(1):E51-60. doi: 10.1002/ccd.25123. Epub 2013 Aug 5. PMID 23832623
- [Background] Duarte PVF, Cortes LA, de Almeida Sampaio FB, Barroso JM, da Silveira GM, Nascif GB, Filho AO, Ribeiro ML, Salles MM, De Lorenzo A. Feasibility and Safety of Ipsilateral Ulnar Access in Cases of Impossibility or Failure of Radial Access for Coronary Angiography or Percutaneous Coronary Intervention. J Invasive Cardiol. 2022 Feb;34(2):E92-E97. doi: 10.25270/jic/21.00138. Epub 2022 Jan 16. PMID 35037897
- [Background] Bernat I, Aminian A, Pancholy S, Mamas M, Gaudino M, Nolan J, Gilchrist IC, Saito S, Hahalis GN, Ziakas A, Louvard Y, Montalescot G, Sgueglia GA, van Leeuwen MAH, Babunashvili AM, Valgimigli M, Rao SV, Bertrand OF; RAO International Group. Best Practices for the Prevention of Radial Artery Occlusion After Transradial Diagnostic Angiography and Intervention: An International Consensus Paper. JACC Cardiovasc Interv. 2019 Nov 25;12(22):2235-2246. doi: 10.1016/j.jcin.2019.07.043. PMID 31753298
- [Background] Hahalis G, Aznaouridis K, Tsigkas G, Davlouros P, Xanthopoulou I, Koutsogiannis N, Koniari I, Leopoulou M, Costerousse O, Tousoulis D, Bertrand OF. Radial Artery and Ulnar Artery Occlusions Following Coronary Procedures and the Impact of Anticoagulation: ARTEMIS (Radial and Ulnar ARTEry Occlusion Meta-AnalysIS) Systematic Review and Meta-Analysis. J Am Heart Assoc. 2017 Aug 23;6(8):e005430. doi: 10.1161/JAHA.116.005430. PMID 28838915
- [Background] Sgueglia GA, Hassan A, Harb S, Ford TJ, Koliastasis L, Milkas A, Zappi DM, Navarro Lecaro A, Ionescu E, Rankin S, Said CF, Kuiper B, Kiemeneij F. International Hand Function Study Following Distal Radial Access: The RATATOUILLE Study. JACC Cardiovasc Interv. 2022 Jun 27;15(12):1205-1215. doi: 10.1016/j.jcin.2022.04.023. Epub 2022 May 17. PMID 35595672
- [Background] Zwaan EM, Cheung ES, IJsselmuiden AJJ, Holtzer CAJ, Schreuders TAR, Kofflard MJM, Coert JH. Upper Extremity Function following Transradial Percutaneous Coronary Intervention: Results of the ARCUS Trial. J Interv Cardiol. 2022 Sep 6;2022:6858962. doi: 10.1155/2022/6858962. eCollection 2022. PMID 36128073
- [Background] Valgimigli M, Campo G, Penzo C, Tebaldi M, Biscaglia S, Ferrari R; RADAR Investigators. Transradial coronary catheterization and intervention across the whole spectrum of Allen test results. J Am Coll Cardiol. 2014 May 13;63(18):1833-41. doi: 10.1016/j.jacc.2013.12.043. Epub 2014 Feb 26. PMID 24583305
- [Background] Kolkailah AA, Alreshq RS, Muhammed AM, Zahran ME, Anas El-Wegoud M, Nabhan AF. Transradial versus transfemoral approach for diagnostic coronary angiography and percutaneous coronary intervention in people with coronary artery disease. Cochrane Database Syst Rev. 2018 Apr 18;4(4):CD012318. doi: 10.1002/14651858.CD012318.pub2. PMID 29665617